CLINICAL TRIAL: NCT04307992
Title: Feasibility Assessment of the Prophylactic Use of AneuFix at the Time of EVAR Implantation
Brief Title: AneuFix - Prophylactic Sac Filling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TripleMed B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Triplemed 003
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Abdominal Aortic Aneurysm; Endoleak
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Intervention Model Description: The current study is a follow-up study on the previous feasibility study where ACP-T5 was used. After increasing the % tantalum in ANEUFIX to make the product more detectable under X-ray, the current study is a pilot study that (1) evaluates the technical feasibility of the prophylactic use of AneuFix during EVAR implentation and (2) assesses the rate of endoleaks after EVAR in 5 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Device: ANEUFIX
  Interventions: Device: Prophylactic sac filling with AneuFix

INTERVENTIONS:
Device: Prophylactic sac filling with AneuFix — ANEUFIX is administered by injection into the AAA via transferal access at the time of EVAR placement using imaging techniques to guide the place of injection.

SUMMARY:
This study is set up to assess the feasibility and safety of the clinical procedure using AneuFix in a prophylactic setting at the time of EVAR endograft implantation.

DETAILED DESCRIPTION:
The investigational device is called ANEUFIX, which is a product treating the endoleak by blockage of backflowing blood vessels, i.e. by filling the endoleak void and nidus of feeding artery and exit of existing draining arteries.

ANEUFIX is a polymer that cures rapidly (2-4 min at 37°C) after injection into the AAA-sac close to the nidus.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic, infrarenal AAA that requires surgery with a high-risk profile of developing endoleak type II in line with the recommendations of Guntner et al:

  - Open IMA AND
  * 1 patent lumbar AND a cross-sectional area at the location of the IMA (CSAIMA) >17,5cm2 OR
  * 2 patent lumbars AND a CSAIMA >15cm2 OR
  * 3 patent lumbars AND a CSAIMA >12,5 cm2 OR
  * 4 patent lumbars AND a CSAIMA >10 cm2 OR
  * 5 patent lumbars AND a CSAIMA >7,5 cm2
* Infrarenal neck according to the IFU of the EVAR device
* Other aortic-iliac anatomical configuration suitable for EVAR according to the criteria of the EVAR device to be used
* Patient having a life expectation of at least 2 years
* Being older than 18 years
* Willing and able to comply with the requirements of this clinical study

Exclusion Criteria:

* Patient not able or willing to give written Informed Consent
* Patient undergoing emergency procedures
* Patient undergoing EVAR for ruptured or symptomatic AAA,
* Patient with a suprarenal AAA
* Patient with an inflammatory AAA (more than minimal wall thickening)
* Patient with an infrarenal neck unsuitable for endovascular fixation (including so called "hostile necks") or aortic-iliac anatomic configuration otherwise unsuitable for EVAR according to criteria of the device to be used
* Patient in which a bilateral retroperitoneal incision is required for EVAR
* Patient in which a sacrifice of both hypogastric arteries is required
* Patient with anatomical variations, i.e. horseshoe-kidney, arteries requiring reimplantation
* Patient in which the administration of contrast agent is not possible: proved, severe systemic reaction to contrast agent
* Patient with active infection present
* Patients scheduled for or having received an organ transplant
* Patient with limited life expectation due to other illness (<1 year)
* Patient with non-iatrogenic bleeding diathesis
* Patient with connective tissue disease
* Women of child-bearing potential
* Patients with evidence at completion angiogram during EVAR of a type Ia or type III endoleak persistent after balloon inflation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical Success | 24 hours
  Technical Success as demonstrated by the feasibility to fill the AAA sac after EVAR during the same procedure, and by the rate of (all) endoleaks after EVAR followed by the AneuFix procedure
Clinical Success rate | 6 months
  Clinical Success as demonstrated by the occurrence of type II endoleaks at 6 months after EVAR, and aneurysmal sac growth at 6 months after EVAR
Clinical Success rate | 12 months
  Clinical Success as demonstrated by the occurrence of type II endoleaks at 12 months after EVAR, and aneurysmal sac growth at 12 months after EVAR

SECONDARY OUTCOMES:
Intraoperative occurrence of complications | 24 hours
  Adverse events occurring during the surgical intervention are registered.
Peri-operative complications | 30 days
  Rate of peri-operative complications
Prevention of (any type of) endoleak | 1, 6 and 12 months
  Occurrence of (any type of) endoleak
adverse events | 1, 6 and 12 months
  Occurrence of adverse events and adverse device effects
Re-interventions | 1, 6 and 12 months
  Rate of secondary endovascular or surgical re-interventions
Aneurysm rupture | 6 and 12 months
  Rate of aneurysm rupture
Proportion of patients surviving 24 months after treatment | 24 months
  Survival throughout the study up until 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Arjan WJ Hoksbergen, Dr, Principal Investigator — VUmc Heelkunde, Amsterdam
Locations (1):
- VUmc, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Smorenburg SPM, Lely RJ, Jongkind V, Groeneveld ME, de Vries AC, Brom HLF, Jacobs MJ, Hoksbergen AWJ. First in Human Aortic Aneurysm Sac Filling with AneuFix Injectable Polymer during Endovascular Aneurysm Repair. Eur J Vasc Endovasc Surg. 2025 Dec 29:S1078-5884(25)01317-6. doi: 10.1016/j.ejvs.2025.12.048. Online ahead of print. PMID 41475431
- [Derived] Smorenburg SPM, Lely RJ, Jacobs MJ, Hoksbergen AWJ. Aortic aneurysm sac filling with AneuFix injectable polymer during endovascular aneurysm repair: feasibility and safety trial study protocol. BMJ Open. 2024 Jul 15;14(7):e082380. doi: 10.1136/bmjopen-2023-082380. PMID 39009453